CLINICAL TRIAL: NCT01242202
Title: Phase III Study of ASP1941 - Open-label, Non-comparative Study to Assess the Long-term Safety, Tolerability and Efficacy of ASP1941 in Combination With an α-Glucosidase Inhibitor in Japanese Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control With an α-Glucosidase Inhibitor Alone
Brief Title: A Study to Assess the Safety and Efficacy of ASP1941 in Combination With α-glucosidase Inhibitor in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1941-CL-0108
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes mellitus; alpha glucosidase inhibitor; ASP1941; long-term safety
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ipragliflozin; Glycoside Hydrolase Inhibitors; Acarbose; miglitol; voglibose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP group (Experimental): Concomitant administration of ASP1941 and α- glucosidase inhibitor
  Interventions: Drug: ipragliflozin; Drug: alpha glucosidase inhibitor

INTERVENTIONS:
Drug: ipragliflozin — oral
  Other Names: ASP1941
Drug: alpha glucosidase inhibitor — oral
  Other Names: Acarbose; Miglitol; Voglibose

SUMMARY:
This study is to evaluate long-term safety and efficacy after concomitant administration of ASP1941 and α-glucosidase inhibitor in Japanese patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a 52-week multi-center study in subjects with type 2 diabetes mellitus who have inadequate glycemic control on an α-Glucosidase Inhibitor alone. Dosage may be increased during the treatment period if subjects fulfill increasing criteria and the investigators adjudicate that no impact for subjects safety.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients receiving with α-glucosidase inhibitor mono-therapy for at least 4 weeks
* HbA1c value between 6.5 and 9.5%
* Body Mass Index (BMI) 20.0 - 45.0 kg/m2

Exclusion Criteria:

* Type 1 diabetes mellitus patients
* Serum creatinine > upper limit of normal
* Proteinuria (albumin/creatinine ratio > 300mg/g)
* Dysuria and/or urinary tract infection, genital infection
* Significant renal, hepatic or cardiovascular diseases
* Severe gastrointestinal diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2010-10-21 (Actual); Primary Completion 2012-05-25 (Actual); Study Completion 2012-05-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | baseline and 52 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose | baseline and 52 weeks
Change from baseline in fasting serum insulin | baseline and 52 weeks
Safety as reflected by adverse events, routine safety laboratories, vital signs, physical examinations and 12-lead electrocardiograms (ECGs) | for 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (6):
- Japan (6):
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=102